CLINICAL TRIAL: NCT04998877
Title: Physical Activity, Cardiac and Skeletal Muscle Energetics in Healthy Subjects and HFpEF Patients
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00270339
Record Dates: First submitted 2021-07-28; First posted 2021-08-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure with Preserved Ejection Fraction
- Healthy Volunteers

SUMMARY:
This research is being done to better understand the relationship between information collected by wearable devices and clinical measurements in people with heart failure with preserved ejection fraction (HFpEF) and others without HFpEF. This is an observational study with no study intervention or randomization.

Participants will undergo baseline history and physical, 12-lead EKG, laboratory studies of blood/serum/urine, echocardiography, activity questionnaire, 6 minute walk test, and placement of wearable devices to be worn for up to 14 days (activity monitors, EKG monitor and continuous glucose monitor).

Participants will return after ~14 days of wearing the devices and repeat of physical examination, 12-lead EKG, 6 minute walk test, activity questionnaire. Additionally, participants will undergo magnetic resonance imaging (MRI) of their leg with exercise, cardiopulmonary exercise testing (CPET) and, for those who qualify, magnetic resonance imaging (MRI) of their heart with exercise.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Women and men between the ages of 40 and 85 years, inclusive, at the Screening visit.
* Women of childbearing potential require a negative pregnancy test.
* Participants who are willing and able to comply with all scheduled visits, laboratory tests, lifestyle considerations, and other study procedures.
* Capable of giving signed informed consent, which includes willingness to be compliant with the requirements and restrictions listed in the informed consent document and in this protocol.

Healthy Participants Only :

* Healthy participants with no history of diabetes mellitus, or significant heart or vascular disease, including a history of heart failure, myocardial infarction, revascularization or positive exercise tolerance test for ischemia (if previously performed).
* BMI of 30.0 - 50.0 kg/m2, inclusive

Heart Failure Participants Only:

* Previous clinical diagnosis of heart failure with New York Heart Association (NYHA) Class II-IV symptoms at screening visit and present for at least 1 month.
* Symptom(s) of HF requiring treatment with diuretic(s) for at least 30 days prior to screening
* Left ventricular ejection fraction (EF) >=50% by echocardiography, MRI, CT or x-ray or nuclear ventriculography at screening visit or within prior 12 months.
* Patients with at least 1 of the following:
* HF hospitalization (defined as HF listed as the major reason for hospitalization and treatment with diuretics) or outpatient diuresis visit within 24 months prior to screening visit OR
* evidence of structural cardiac changes or elevated biomarkers. The structural changes are defined by at least 1 of the following echocardiography findings (any local measurement made during the screening epoch or within the 6 months prior to screening visit):
* Left Atrium (LA) enlargement defined by at least 1 of the following: LA width (diameter) ≥3.8 cm or LA length ≥5.0 cm or LA area ≥20 cm2 or LA volume ≥55 ml or LA volume index ≥29 ml/m2 ,
* Left Ventricular Hypertrophy (LVH) defined by septal thickness or posterior wall thickness ≥1.1 cm.
* The biomarker changes are defined as N terminal (NT)-proBNP >200 pg/ml for patients not in atrial fibrillation (AF) or >600 pg/ml for patients in AF on screening.
* Stable cardiovascular medical therapy for at least 30 days, defined as no addition or removal or major (>100%) dose change of prescribed medications for the treatment of cardiovascular disease such as, but not limited to: Renin-Angiotensin-Aldosterone System (RAAS) antagonists, beta-blockers, or calcium channel blockers for hypertension.
* At Visit 1 (Screen 1), BMI of 30.0 - 50.0 kg/m2, inclusive.

Exclusion Criteria:

All participants

Participants are excluded from the study if any of the following criteria apply:

* Age < 40 years or > 85 years
* A history of myocardial infarction, stroke, or transient ischemic attack, within 6 months of Screen 1 (Visit 1);
* Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin); a subject is considered cured if there has been no evidence of cancer recurrence in the previous 5 years.
* Participants with any contraindication to MRI scanning or an anatomical or pathological abnormality that would either preclude or tend to confound the analysis of study data, including the following:
* History of severe claustrophobia impacting ability to perform MRI during the study
* Implanted metallic objects contraindicated in MRI such as (pre-existing cardiac pacemakers, cerebral clips) or indwelling metallic projectiles;
* Participants unable to fit within MRI scanner or follow instructions.
* Fasting serum triglycerides ≥500 mg/dL (5.6 mmol/L) on current medications
* Fasting LDL-C ≥190 mg/dL (4.9 mmol/L) on current medications

Prior/Concomitant Therapy:

* Use of prior/concomitant weight loss pharmacotherapy or weight loss surgery within the prior six months.

Healthy [Non-HFpEF] Participants Only:

In addition, Healthy Participants presenting with any of the following will not be included in the study:

* Screening supine 12 lead ECG demonstrating evidence of prior infarction or ischemia, significant arrhythmia or clinically significant conduction abnormalities.
* Uncontrolled hypertension, or those participants requiring greater than 2 blood pressure lowering medications.
* Screening Fasting glucose level of ≥126 mg/dL.
* History of diabetes mellitus
* Significant heart or vascular disease, including a history of heart failure, myocardial infarction, revascularization or positive exercise tolerance test for ischemia (if previously performed).
* Other medical or psychiatric condition that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Heart Failure Participants Only:

* History of infiltrative cardiomyopathy or constrictive pericarditis, cor pulmonale, or significant pulmonary disease.
* Significant valvular abnormalities.
* History of clinical coronary artery disease (CAD) or significant epicardial coronary disease (>50% stenosis) in major coronary artery by x-ray or CT angiography unless (a) the patient underwent prior successful revascularization with percutaneous coronary angioplasty within the prior three years.
* Any condition other than HF which could limit the ability to perform a six minute walk test (6MWT) or CPET test (e.g., critical peripheral vascular disease, significant orthopedic or neurological conditions),
* Any diseases other than HF which are likely to significantly alter the patient's global perception of status or quality of life over a period of 6 months.
* Participants who have previously had a transplanted kidney, liver, or heart.
* At Screening, persistent severe, uncontrolled hypertension; for example: seated systolic blood pressure (SBP) ≥180 mm Hg and/or diastolic blood pressure (DBP) ≥105 mm Hg after ≥5 minute of seated rest, with a single repeat permitted to assess eligibility, if needed.
* At Screening, participants with an estimated glomerular filtration rate (eGFR) of ≤30 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, and serum creatinine (SCr).
* Patients taking combined glucagon-like peptide and gastric inhibitory polypeptide (GLP-1/GIP) receptor agonists at the time of the screening study visit.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are clinical patients of Johns Hopkins or an affiliate of Johns Hopkins.
  Individuals who are clinical patients of the PI or co-investigators. Individuals who are not clinical patients of the PI or coinvestigators. Referral of individuals specifically for research purposes by treating clinicians not on the study team Prior Hopkins/Affiliates study participants Individuals who learn about the study through advertisements or peer/network recruiting
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference of daily activity measures based on accelerometry between HFpEF participants and adults without HFpEF. | Up to 28 days
  Moderate to Vigorous Physical Activity (MVPA; minutes per day); Non-sedentary activity (i.e. sum of light activity and MVPA minutes per day.

SECONDARY OUTCOMES:
Difference of additional daily activity measures based on accelerometry between HFpEF participants and adults without HFpEF. | Up to 28 days
  Sedentary Activity (minutes per day);
Rate of skeletal muscle phosphocreatine (PCr) decline during exercise normalized by work performed. | Up to 28 days
  Difference between adults with and without HFpEF in rate of skeletal muscle [PCr] decline during exercise normalized by work performed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hosptial, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No